CLINICAL TRIAL: NCT00429897
Title: Double Blind Crossover Comparison od Diuretics in Young Patients With Low Renin Hypertension
Brief Title: Double Blind Crossover Comparison of Diuretics in the Young
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Cambridge (Other)
Collaborators: British Heart Foundation (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1.0
Record Dates: First submitted 2007-01-31; First posted 2007-02-01 (Estimated); Last update posted 2007-02-01 (Estimated); Status verified 2007-01

CONDITIONS: Low-Renin Hypertension
Keywords: Hypertension; Low Renin
MeSH Terms: conditions — Hypertension | interventions — Bendroflumethiazide; Amiloride; Spironolactone; Furosemide

INTERVENTIONS:
Drug: Bendroflumethiazide 2.5mg - 5mg
Drug: Amiloride 20-40mg
Drug: Spironolactone 50-100mg
Drug: Frusemide 20-40mg
Drug: Bendroflumethiazide 1.25-2.5mg/ Amiloride 10-20mg combined

SUMMARY:
The principle objective of the study is to determine whether low-renin (i.e. salt sensitive) hypertension at a young age is caused by the kidneys hanging onto too much salt as a result of an over active salt pump in the kidney.

The kidneys have four different salt pumps, and each is blocked by a different type of diuretic (salt losing tablet)If one out of the four is overactive, we would expect patients to respond much better to one diuretic than to the alternatives - rather than responding equally well to all available types of diuretic.

DETAILED DESCRIPTION:
Studies suggest that patients with low renin hypertension respond better to diuretics than other hypertensive drug groups. The aim of the study is to rotate patients through the four main diuretic groups and see if it is possible to identify the most effective diuretic for this group, as measured by a >=10mgHg decrease in Systolic blood pressure in one specific group a compared to the others.

As most caucasians with Low renin hypertension are older (>55), presentation with this type of hypertension at a younger age suggests the presence of substantial genetic variation in order to cause the atypical presentation. It is hoped that by identifying the best diuretic for these patients we will also be able to identify:

1. Whether the young low-renin hypertensives can be sub-classified according to their most effective diuretic;
2. Whether this sub-classification helps us to identify the genes and mutations responsible, since these are to expected to be in the so-called sodium channels (i.e. salt pumps)which the kidneys use to prevent salt being excreted in the urine.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-45
* male or female
* Hypertensive - 3 clinic SBP >=140mmHg; or 3 clinic DBP >=90mmHg; or ABPM or home BP >=130(SBP) or 85(DBP)
* 24hr Na+<160mmol/l
* EITHER {Plasma renin<=10mU/L (measured untreated, or whilst receiving only CCB+/-diuretic} + {Plasma renin <=40mU/L (measured on an ACEi or ARB, which approximately double s the plasma renin)} OR Plasma renin <5mU/L (measured untreated, or receiving any antihypertensive drug other than a beta-blocker

Exclusion Criteria:

* Documented history of gout
* Abnormal renal function (both elevated serum creatinine and reduced creatinine clearance
* SBP > 170mmHg or Diastolic >110mmHg despite treatment with permitted background treatment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30
Dates: Start 2006-08; Study Completion 2007-07

PRIMARY OUTCOMES:
Difference in systolic blood pressure for subjects' best drug and second best drug.
Difference in plasma renin for subjects' best drug and second best drug.

SECONDARY OUTCOMES:
Predictions of best drug

CONTACTS AND LOCATIONS:
Overall Officials: Morris J Brown, Proffessor, Principal Investigator — Cambridge University
Locations (1):
- University of Cambridge - Addenbrookes Hospital, Cambridge, United Kingdom